CLINICAL TRIAL: NCT03304379
Title: Phase 3 Randomized, Double-Blind, Multi-Dose, Placebo And NSAID Controlled Study To Evaluate The Efficacy And Safety Of Fasinumab In Patients With Pain Due To Osteoarthritis Of The Knee Or Hip
Brief Title: Study to Determine the Safety and the Efficacy of Fasinumab Compared to Placebo and Nonsteroidal Anti-inflammatory Drugs (NSAIDs) for Treatment of Adults With Pain From Osteoarthritis of the Knee or Hip
Acronym: FACT OA2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R475-OA-1688; 2017-001702-15 (EudraCT Number)
Record Dates: First submitted 2017-10-02; First posted 2017-10-09 (Actual); Results first posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — fasinumab; Diclofenac; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dosing regimen 1 (Experimental)
  Interventions: Drug: Fasinumab; Drug: Matching placebo
- Dosing regimen 2 (Experimental)
  Interventions: Other: Diclofenac; Drug: Matching placebo
- Dosing regimen 3 (Experimental)
  Interventions: Other: Celecoxib; Drug: Matching placebo
- Dosing regimen 4 (Experimental)
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Fasinumab — Solution for injection in pre-filled syringe
  Other Names: REGN475; MT-5547
  Arms: Dosing regimen 1
Other: Diclofenac — NSAID active comparator (capsule)
  Other Names: ZORVOLEX
  Arms: Dosing regimen 2
Other: Celecoxib — NSAID active comparator (capsule)
  Other Names: CELEBREX
  Arms: Dosing regimen 3
Drug: Matching placebo — Fasinumab-matching placebo (solution for injection in pre-filled syringe); NSAID-matching placebo (capsule)

SUMMARY:
The primary objective of the study is to evaluate the efficacy of fasinumab compared to placebo, when administered for up to 24 weeks in patients with pain due to osteoarthritis (OA) of the knee or hip.

The secondary objectives of the study are:

* To evaluate the efficacy of fasinumab compared to non-steroidal anti-inflammatory drugs (NSAID)s, when administered for up to 24 weeks in patients with pain due to OA of the knee or hip
* To assess the safety and tolerability of fasinumab compared to placebo and compared to NSAIDs, when administered for up to 24 weeks in patients with pain due to OA of the knee or hip

ELIGIBILITY:
Key Inclusion Criteria (additional criteria may apply at screening):

1. A clinical diagnosis of osteoarthritis (OA) of the knee or hip based on the American College of Rheumatology criteria with radiologic evidence of OA (K-L score ≥2 for the index joint) at the screening visit.
2. Willing to discontinue current pain medications and to adhere to study requirements for rescue treatments (acetaminophen/paracetamol to be taken as needed with a maximum daily dose of 2500 mg [countries where 500 mg strength tablets/capsules are available] or 2600 mg [countries where 325 mg strength tablets/capsules are available])
3. A history of at least 12 weeks of inadequate pain relief or intolerance to analgesics used for pain due to OA of the knee or hip
4. Currently using a stable dose of NSAID
5. Willing to discontinue glucosamine sulfate and chondroitin sulfate treatments during the 24 weeks of treatment

Key Exclusion Criteria (additional criteria may apply at screening):

1. Non-compliance with the numeric rating scale (NRS) recording during the pre-randomization period
2. History or presence at the screening visit of non-OA inflammatory joint disease, Paget's disease of the spine, pelvis or femur, neuropathic disorders, multiple sclerosis, fibromyalgia, tumors or infections of the spinal cord, or renal osteodystrophy
3. History or presence on imaging of arthropathy, hip or knee dislocation, extensive subchondral cysts, evidence of severe structural damage, bone collapse, or primary metastatic tumor with the exception of chondromas or pathologic fractures
4. Trauma to the index joint within 3 months prior to the screening visit
5. Signs or symptoms of carpal tunnel syndrome within 6 months of screening
6. Patient is not a candidate for magnetic resonance imaging (MRI)
7. Is scheduled for a JR surgery to be performed during the study period or who would be unwilling or unable to undergo JR surgery if needed
8. History or presence at the screening visit of autonomic or diabetic neuropathy, or other peripheral neuropathy, including reflex sympathetic dystrophy
9. Evidence of autonomic neuropathy as defined in the schedule of assessments (SoAs)
10. History or diagnosis of chronic autonomic failure syndrome including pure autonomic failure, multiple system atrophy
11. Use of systemic corticosteroids within 30 days prior to the screening visit. Intra-articular corticosteroids in the index joint within 12 weeks prior to the screening visit, or to any other joint within 30 days prior to the screening visit
12. Exposure to an anti-NGF antibody prior to the screening visit or known sensitivity or intolerance to anti-NGF antibodies
13. Women of childbearing potential who are unwilling to practice highly effective contraception prior to the start of the first treatment, during the study, and for at least 20 weeks after the last dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1650 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (71):
- United States (71):
  - Pinnacle Research Group, Llc, Anniston, Alabama
  - Horizon Research Partners, Mobile, Alabama
  - Clinical Research Advantage, Inc./Warner Family Practice, PC, Chandler, Arizona
  - Synexus Central Phoenix Medical Clinic, Phoenix, Arizona
  - Clinical Research Consortium Arizona, Tempe, Arizona
  - Advance Research Center, Anaheim, California
  - TriWest Research Associates, LLC, El Cajon, California
  - Paragon Rx Clinical Research, Inc., Garden Grove, California
  - Catalina Research Institute, LLC, Montclair, California
  - Sierra Clinical Research, Roseville, California
  - UC Davis Center for Musculoskeletal Health, Sacramento, California
  - Advanced Research Center, Inc, San Diego, California
  - California Research Foundation, San Diego, California
  - Paragon Rx Clinical Research, Inc, Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - Westlake Medical Research, Thousand Oaks, California
  - Synexus Clinical Research US, Inc., Vista, California
  - Mountain View Clinical Research, Denver, Colorado
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - CRM of Greater New Haven, LLC, Hamden, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Avail Clinical Research, LLC, DeLand, Florida
  - AMB Research Center, Inc, Miami, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - Lakes Research, LLC, Miami Lakes, Florida
  - Bioclinica Research, Orlando, Florida
  - Gulf Region Clinical Research institute, Pensacola, Florida
  - Integral Rheumatology & Immunology Specialists (IRIS), Plantation, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Drug Studies America, Marietta, Georgia
  - Georgia Institute For Clinical Research LLC, Marietta, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Chicago Clinical Research Institute, Inc, Chicago, Illinois
  - Affinity Clinical Research Institute, Oak Lawn, Illinois
  - Clinical Research Advantage, Inc., Evansville, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - L-MARC Research Center, Louisville, Kentucky
  - Tandem Clinical Research, Marrero, Louisiana
  - Tufts Medical Center, Inc., Boston, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Onyx Clinical Research, Caro, Michigan
  - Synexus Clinical Research US, Inc., Richfield, Minnesota
  - Skyline Medical Center /Radiant Research, Inc., Elkhorn, Nebraska
  - Meridian Clinical Research Associates, LLC, Omaha, Nebraska
  - Robert Kaplan, D.O., Las Vegas, Nevada
  - Amici Clinical Research, LLC, Raritan, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Drug Trial Brooklyn, Brooklyn, New York
  - Northwell Health, Great Neck, New York
  - Drug Trials America, Hartsdale, New York
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - Carolina Research Center, Shelby, North Carolina
  - PMG Research of Wilmington LLC, Wilmington, North Carolina
  - The Center For Clinical Research, Winston-Salem, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Aventiv Research Inc, Columbus, Ohio
  - DOC Clinical Research, Dayton, Ohio
  - Center for Orthopaedics and Sports Medicine, Indiana, Pennsylvania
  - Radiant Research, Inc., Anderson, South Carolina
  - Piedmont Comprehensive Pain Management Group, Greenville, South Carolina
  - Radiant Research, Inc., Greer, South Carolina
  - Coastal Carolina Research Center at LowCountry Orthopaedics, North Charleston, South Carolina
  - Piedmont Research Partners, LLC, Old Point Station, South Carolina
  - ACME Research, LLC, Orangeburg, South Carolina
  - Office of Dr.Ramesh C. Gupta MD, Memphis, Tennessee
  - West Texas Clinical Research, Lubbock, Texas
  - Clinical Investigations Of Texas, Plano, Texas
  - Synexus USA, Plano, Texas
  - Charlottesville Medical Research Center LLC, Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc, Newport News, Virginia
  - Spokane Joint Replacement Center, Spokane, Washington

REFERENCES:
- [Derived] DiMartino SJ, Gao H, Eng S, Valenzuela G, Fuerst T, Emeremni C, Ho T, Hassan HE, Turner KC, Davis JD, Zaim S, Chao J, Patel Y, Brener L, Trinh N, Manvelian G, Fetell M, Braunstein N, Geba GP, Dakin P. Efficacy and safety of fasinumab in an NSAID-controlled study in patients with pain due to osteoarthritis of the knee or hip. BMC Musculoskelet Disord. 2025 Feb 25;26(1):192. doi: 10.1186/s12891-025-08402-8. PMID 40001000

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 4531 participants were screened in this study. Out of which, 1650 participants were randomized to 1 of the following arms: Fasinumab (1 milligram [mg]), non-steroidal anti-inflammatory drug (NSAIDs), matched placebo, Fasinumab 3 and 6 mg. Screen failure was mostly due to inclusion criteria not met/exclusion criteria met. Eligible participants were randomized to receive placebo matched to Fasinumab/NSAIDs, NSAIDs (Diclofenac and Celecoxib) and Fasinumab 1 mg.
Pre-assignment Details: In May 2018, the sponsor implemented an urgent safety measure to stop dosing for participants randomized to Fasinumab (6 mg and 3 mg), to prevent further randomization to these regimens across the Fasinumab program based on review of unblinded data in an ongoing study R475-PN-1523 (NCT02683239). Participants from Fasinumab 3 mg and 6 mg group were moved directly into the 20-week follow-up period.
Groups:
- Placebo: Participants who received subcutaneous (SC) injection of placebo matched to Fasinumab every 4 weeks (Q4W) or every 8 weeks (Q8W) alternatively or oral placebo matched to NSAID twice daily (BID) up to 24 weeks.
- NSAIDs: Participants received oral capsule of Diclofenac at a dose of 75 mg BID or oral capsule of Celecoxib at a dose of 200 mg once daily (QD) up to 24 weeks.
- Fasinumab 1 mg: Participants received SC injection of Fasinumab at a dose of 1 mg Q4W up to 24 weeks and NSAID-matching placebo oral, BID
- Fasinumab 3 mg: Participants received SC injection of Fasinumab at a dose of 3 mg Q4W up to 24 weeks and NSAID-matching placebo oral, BID
- Fasinumab 6 mg: Participants received SC injection of Fasinumab at a dose of 6 mg Q8W up to 24 weeks, alternating with Q8W placebo injections. Participants received placebo injections at the Q4W study visits where study drug was not administered and NSAID-matching placebo oral, BID
Period: Overall Study
Arm/Group | Placebo | NSAIDs | Fasinumab 1 mg | Fasinumab 3 mg | Fasinumab 6 mg
Started | 308 | 612 | 612 | 59 | 59
Full Analysis Set (FAS) (FAS included all randomized participants excluding participants affected by the urgent safety measure and was based on the treatment allocated (as randomized)) | 308 | 612 | 612 | 0 | 0
Safety Analysis Set (SAF) (SAF included all randomized participants from the FAS who received any study drug. It is based on the actual treatment received.) | 309 | 609 | 609 | 0 | 0
Urgent Safety Measure Set (USMS) (USMS included all participants randomized to Fasinumab 3 mg Q4W or 6 mg Q8W and was based on the treatment allocated (as randomized)) | 0 | 0 | 0 | 59 | 59
Completed Treatment | 218 | 436 | 454 | 0 | 0
Completed | 238 | 471 | 463 | 42 | 42
Not Completed | 70 | 141 | 149 | 17 | 17
Not completed — Protocol Violation | 8 | 10 | 5 | 0 | 2
Not completed — Adverse Event | 4 | 20 | 17 | 1 | 0
Not completed — Lack of Efficacy | 17 | 16 | 20 | 0 | 0
Not completed — Physician Decision | 6 | 10 | 6 | 9 | 10
Not completed — Withdrawal by Subject | 26 | 58 | 66 | 3 | 5
Not completed — Lost to Follow-up | 8 | 24 | 35 | 4 | 0
Not completed — Death | 1 | 2 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | NSAIDs | Fasinumab 1 mg | Fasinumab 3 mg | Fasinumab 6 mg | Total
Number analyzed (Participants) | 308 | 612 | 612 | 59 | 59 | 1650
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (9.30) | 62.3 (9.41) | 62.1 (9.13) | 62.8 (9.38) | 61.5 (9.55) | 62.2 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 418 | 436 | 36 | 34 | 1146
  Male | 86 | 194 | 176 | 23 | 25 | 504
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 44 | 31 | 5 | 10 | 110
  Not Hispanic or Latino | 285 | 568 | 581 | 54 | 49 | 1537
  Unknown or Not Reported | 3 | 0 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 0 | 2
  Asian | 33 | 57 | 54 | 8 | 3 | 155
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 0 | 2
  Black or African American | 60 | 134 | 132 | 12 | 16 | 354
  White | 202 | 396 | 405 | 39 | 40 | 1082
  More than one race | 11 | 24 | 18 | 0 | 0 | 53
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 2
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score [Mean (Standard Deviation); unit: Score on a scale] — WOMAC pain subscale was a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index joint (knee or hip) in the past 48 hours. It was calculated as the mean of the scores from the 5 individual questions scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (higher pain), where higher scores indicated higher pain. Population: Here 'n' = number of evaluable participants at the specified time point
  Score on a scale
    number analyzed (Participants) | 308 | 611 | 612 | 58 | 59 | 1648
    (all) | 6.42 (1.394) | 6.38 (1.344) | 6.46 (1.321) | 6.43 (1.401) | 6.54 (1.279) | 6.42 (1.344)
WOMAC Physical Function Subscale Scores [Mean (Standard Deviation); unit: Score on a scale] — WOMAC physical function subscale:17-item questionnaire used to assess degree of difficulty experienced due to OA in index joint during past 48 hours. It was calculated as mean of scores from 17 individual questions scored on a NRS of 0 (minimum difficulty) to 10 (maximum difficulty), where higher scores indicated maximum difficulty. Population: Here 'n' = number of evaluable participants at the specified time point
  Score on a scale
    number analyzed (Participants) | 304 | 609 | 610 | 58 | 57 | 1638
    (all) | 6.40 (1.495) | 6.32 (1.418) | 6.39 (1.462) | 6.50 (1.350) | 6.34 (1.392) | 6.37 (1.445)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Scores up to Week 24 in Participants Treated With Fasinumab Compared to Placebo
Description: WOMAC pain subscale was a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index joint (knee or hip) in past 48 hours. It was calculated as the mean of the scores from the 5 individual questions scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (higher pain), where higher scores indicated higher pain.
Time Frame: Baseline up to Week 24
Population: This outcome measure examined only placebo vs. fasinumab 1mg arms. Here, "Number of Subjects Analysed" signifies those subjects who were evaluable for this endpoint. Modified full analysis set (mFAS) includes all randomized participants in FAS but excludes participants from 4 sites for which there were potential concerns regarding data quality, identified prior to database lock.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fasinumab 1 mg
Number analyzed (Participants) | 208 | 439
Score on a Scale
  FAS | -2.21 (0.165) | -2.84 (0.127)
  mFAS: number analyzed (Participants) | 173 | 372
  mFAS | -2.01 (0.182) | -2.78 (0.141)
Statistical Analysis 1: Comparison: Placebo vs Fasinumab 1 mg; Analyses were based on a multiple imputation approach using a Mixed-Effect Model With Repeated Measure (MMRM) model with baseline randomization strata, baseline, treatment, visit and treatment by-visit interaction; Test type: Superiority; p = 0.0003, MMRM — Threshold for significance at 0.05 level; Least Square (LS) Mean Difference = -0.63, 95% CI 2-sided [-0.971 to -0.286]
Statistical Analysis 2: Comparison: Placebo vs Fasinumab 1 mg; (mFAS) Analyses were based on a multiple imputation approach using a MMRM model with baseline, randomization strata, baseline, treatment, visit and treatment by-visit interaction; Test type: Superiority; p > 0.0001, MMRM — Threshold for significance at 0.05 level; LS Mean Difference = -0.77, 95% CI 2-sided [-1.154 to -0.383]

2. Primary Outcome: Change From Baseline in WOMAC Physical Function Subscale Scores up to Week 24 in Participants Treated With Fasinumab Compared to Placebo
Description: Physical function referred to participant's ability to move around and perform usual activities of daily living. The WOMAC physical function subscale was a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in index joint (knee or hip) during past 48 hours. It was calculated as mean of the scores from 17 individual questions scored on a NRS of 0 (minimum difficulty) to 10 (maximum difficulty), where higher scores indicated maximum difficulty.
Time Frame: Baseline up to Week 24
Population: This outcome measure examined only placebo vs. fasinumab 1mg arms. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this endpoint. The modified full analysis set (mFAS) includes all randomized participants in the FAS but excludes participants from four sites for which there were potential concerns regarding data quality, identified prior to database lock.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fasinumab 1 mg
Number analyzed (Participants) | 208 | 439
Score on a Scale
  FAS: number analyzed (Participants) | 207 | 439
  FAS | -2.02 (0.164) | -2.65 (0.125)
  mFAS: number analyzed (Participants) | 172 | 372
  mFAS | -1.80 (0.180) | -2.62 (0.138)
Statistical Analysis 1: Comparison: Placebo vs Fasinumab 1 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0003, MMRM — Threshold for significance at 0.05 level; LS Mean Difference = -0.64, 95% CI 2-sided [-0.981 to -0.290]
Statistical Analysis 2: Comparison: Placebo vs Fasinumab 1 mg; (mFAS) Analyses were based on a multiple imputation approach using an Mixed-Effect Model With Repeated Measure (MMRM) model with baseline randomization strata, baseline, treatment, visit and treatment by-visit interaction; Test type: Superiority; p < 0.0001, MMRM — Threshold for significance at 0.05 level; LS Mean Difference = -0.82, 95% CI 2-sided [-1.198 to -0.443]

3. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (≥) 30 Percent (%) Reduction From Baseline up to Week 24 in WOMAC Pain Subscale Score in Participants Treated With Fasinumab Compared to Placebo
Description: WOMAC pain subscale was a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index knee during past 48 hours. It was calculated as mean of the scores from 5 individual questions scored on a NRS of 0 (minimum pain) to 10 (maximum pain), where higher scores indicate more pain.
Time Frame: Baseline up to Week 24
Population: The FAS included all randomized participants excluding participants affected by the urgent safety measure and was based on the treatment allocated (as randomized). As pre-specified in the protocol, efficacy data from participants randomized to Fasinumab 1 mg Q4W and placebo was only included in the analysis for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Fasinumab 1 mg
Number analyzed (Participants) | 308 | 612
Percentage of Participants | 48.7 | 59.8
Statistical Analysis 1: Comparison: Placebo vs Fasinumab 1 mg; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at 0.05 level. Analyses are based on Cochran-Mantel-Haenszel model; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.581, 95% CI 2-sided [1.195 to 2.092]

4. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) Score up to Week 24 in Participants Treated With Fasinumab Compared to Placebo
Description: The PGA was a patient-rated assessment of current disease state on a 5-point Likert scale where 1 = very good (asymptomatic and no limitation of normal activities), 2 = good (mild symptoms and no limitation of normal activities), 3 = fair (moderate symptoms and limitation of some normal activities), 4 = poor (Severe symptoms and inability to carry out most normal activities) and, 5 =very poor (Very severe symptoms which were intolerable and inability to carry out all normal activities). Higher score indicated severe condition.
Time Frame: Baseline up to Week 24
Population: This outcome measure examined only placebo vs. fasinumab 1mg arms. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this endpoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fasinumab 1 mg
Number analyzed (Participants) | 214 | 440
Score on a Scale | -0.66 (0.063) | -0.81 (0.047)
Statistical Analysis 1: Comparison: Placebo vs Fasinumab 1 mg; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at 0.05 level. Analyses are based on a multiple imputation approach using Mixed-Effect Model With Repeated Measure (MMRM) model; Test type: Superiority; p = 0.0365, MMRM — Threshold for significance at 0.05 level; LS Mean Difference = -0.14, 95% CI 2-sided [-0.28 to -0.009]

5. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Scores up to Week 24 in Participants Treated With Fasinumab Compared to Participants Treated With NSAIDs
Description: WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index joint (knee or hip) in the past 48 hours. It is calculated as the mean of the scores from the 5 individual questions scored on a NRS of 0 (no pain) to 10 (higher pain), where higher scores indicated higher pain.
Time Frame: Baseline up to Week 24
Population: This outcome measure examined only NSAIDs vs. fasinumab 1mg arms. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this endpoint. The modified full analysis set (mFAS) includes all randomized participants in the FAS but excludes participants from four sites for which there were potential concerns regarding data quality, identified prior to database lock.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | NSAIDs | Fasinumab 1 mg
Number analyzed (Participants) | 426 | 439
Score on a Scale
  FAS | -2.60 (0.128) | -2.84 (0.127)
  mFAS: number analyzed (Participants) | 363 | 372
  mFAS | -2.48 (0.140) | -2.78 (0.141)

6. Secondary Outcome: Change From Baseline in WOMAC Physical Function Subscale Scores up to Week 24 in Participants Treated With Fasinumab Compared to Participants Treated With NSAIDs
Description: as for outcome 2
Time Frame: Baseline up to Week 24
Population: This outcome measure examined only NSAIDs vs. fasinumab 1mg arms. Here, "Number of Subjects Analysed" signifies those subjects who were evaluable for this endpoint. The modified full analysis set (mFAS) includes all randomized participants in the FAS but excludes participants from four sites for which there were potential concerns regarding data quality, identified prior to database lock.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | NSAIDs | Fasinumab 1 mg
Number analyzed (Participants) | 426 | 439
Score on a Scale
  FAS | -2.33 (0.127) | -2.65 (0.125)
  mFAS: number analyzed (Participants) | 364 | 372
  mFAS | -2.26 (0.140) | -2.62 (0.138)

7. Secondary Outcome: Change From Baseline in PGA Score up to Week 24 in Participants Treated With Fasinumab Compared to Participants Treated With NSAIDs
Description: as for outcome 4
Time Frame: Baseline up to Week 24
Population: This outcome measure examined only NSAIDs vs. fasinumab 1mg arms. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this endpoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | NSAIDs | Fasinumab 1 mg
Number analyzed (Participants) | 427 | 440
Score on a Scale | -0.75 (0.048) | -0.81 (0.047)

8. Secondary Outcome: Change From Baseline in Weekly Average Walking Index Joint Pain Score up to Week 24 by Using the Numeric Rating Scale (NRS) Pain Scale
Description: Participants reported weekly average walking index joint pain based on NRS. The NRS was nationally recognized numeric scale from 0 to 10, where 0 would demonstrate no pain, 1 to 3 would demonstrate mild pain, 4 to 6 would be moderate pain, 7 to 9 would be severe pain and 10 would be the worst pain possible. Higher score indicated greater pain.
Time Frame: Baseline up to Week 24
Population: This outcome measure examined only placebo, NSAIDs vs. fasinumab 1mg arms. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this endpoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Groups:
- Pooled Placebo: Participants who received subcutaneous (SC) injection of placebo matched to Fasinumab every 4 weeks (Q4W) or every 8 weeks (Q8W) alternatively or oral placebo matched to NSAID twice daily (BID) up to 24 weeks.
Arm/Group | Pooled Placebo | NSAIDs | Fasinumab 1 mg
Number analyzed (Participants) | 231 | 449 | 470
Score on a Scale | -1.85 (0.130) | -2.13 (0.101) | -2.51 (0.100)

9. Secondary Outcome: Number of Participants With Adjudicated Arthropathy (AA) Events
Description: AA was a composite term that encompasses the following conditions: Rapidly progressive Osteoarthritis (OA) type 1 and 2, Subchondral insufficiency fractures, and Primary Osteonecrosis confirmed by an arthropathy adjudication committee. AAs were also evaluated to determine if they met Destructive Arthropathy criteria.
Time Frame: Baseline up to follow-up period (Week 44)
Population: This outcome measure examined only placebo, NSAIDs vs. fasinumab 1mg arms. Safety Analysis set (SAF) included all randomized participants from the FAS who received any study drug. It was based on the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | NSAIDs | Fasinumab 1 mg
Number analyzed (Participants) | 309 | 609 | 609
Participants | 5 | 9 | 34

10. Secondary Outcome: Number of Participants With AA Events Meeting Destructive Arthropathy (DA) Criteria
Description: DA is a unique clinical form of rapidly destructive arthropathy over and above that seen in the normal progression of OA. DA criteria can be associated with Rapidly Progressive OA type 2, Subchondral Insufficiency fracture, and Primary Osteonecrosis confirmed by an arthropathy adjudication committee.
Time Frame: Baseline up to follow-up period (Week 44)
Population: This outcome measure examined only placebo, NSAIDs vs. fasinumab 1mg arms. SAF included all randomized participants from the FAS who received any study drug. It was based on the actual treatment received. Here, "Number of Participants Analyzed" signifies those participants who had positive AA.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | NSAIDs | Fasinumab 1 mg
Number analyzed (Participants) | 5 | 9 | 34
Participants | 0 | 0 | 2

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a study drug which may or may not have a causal relationship with the study drug. TEAE was defined as an AE with an onset that occurs after receiving study drug. A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious TEAEs.
Time Frame: Baseline up to follow-up period (Week 44)
Population: This outcome measure examined only placebo, NSAIDs vs. fasinumab 1mg arms. SAF included all randomized participants from the FAS who received any study drug. It was based on the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | NSAIDs | Fasinumab 1 mg
Number analyzed (Participants) | 309 | 609 | 609
Participants | 186 | 406 | 403

12. Secondary Outcome: Number of Participants With Sympathetic Nervous System (SNS) Dysfunction Events
Description: Potential events of SNS dysfunction were monitored throughout the study through physical examination, AE reporting, assessment of orthostatic hypotension, and the Survey of Autonomic Symptoms. Sympathetic nervous system dysfunction was diagnosed after consultation with an appropriate specialist, such as a neurologist and/or cardiologist.
Time Frame: Baseline up to follow-up period (Week 44)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | NSAIDs | Fasinumab 1 mg
Number analyzed (Participants) | 309 | 609 | 609
Participants | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With At-least One Peripheral Sensory Adverse Events (AEs)
Description: Any participants with a peripheral sensory event that persisted for 2 months was referred for a neurology or other specialty consultation and reported as an Adverse Events of Special Interest (AESI).
Time Frame: Baseline up to Week 44
Population: This outcome measure examined only placebo, NSAIDs vs. fasinumab 1mg arms. SAF included all randomized participants from the FAS who received any study drug. It is based on the actual treatment received
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NSAIDs | Fasinumab 1 mg
Number analyzed (Participants) | 309 | 609 | 609
Participants | 8 | 24 | 31

14. Secondary Outcome: Number of Participants Who Underwent a Joint Replacements (JR) Surgery From Baseline up to Week 24
Description: Number of participants who underwent a JR surgery from baseline up to Week 24 were reported.
Time Frame: Baseline up to Week 24
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NSAIDs | Fasinumab 1 mg
Number analyzed (Participants) | 309 | 609 | 609
Participants | 2 | 7 | 3

15. Secondary Outcome: Number of Participants Who Underwent a Joint Replacements (JR) Surgery From Baseline up to Week 44
Description: Number of participants who underwent a JR surgery from baseline up to follow-up period (Week 44) were reported.
Time Frame: Baseline up to Week 44
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NSAIDs | Fasinumab 1 mg
Number analyzed (Participants) | 309 | 609 | 609
Participants | 6 | 13 | 10

16. Secondary Outcome: Number of Participants With Joint Replacement (JR) Surgery Reported at End of Study (EOS) (Week 72)
Description: An EOS phone contact was conducted at Week 72 following the last dose of study drug (Week 24) to evaluate the number of participants who had undergone or were scheduled for JR surgery.
Time Frame: At Week 72
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NSAIDs | Fasinumab 1 mg
Number analyzed (Participants) | 309 | 609 | 609
Participants | 11 | 29 | 21

17. Secondary Outcome: Serum Concentrations of Functional Fasinumab
Time Frame: At Weeks 0, 4, 8, 16, 24 and 44
Population: Pharmacokinetic (PK) analysis set included all treated participants who received any study drug and who had at least 1 non-missing drug concentration result following the first study dose. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome measure and "Number Analyzed" = participants who were evaluable at specified time points. Data was planned to be collected and analyzed for Fasinumab 1 mg Q4W arm only.
Measure: Mean (Standard Deviation); unit: Milligrams per Liter (mg/L)
Arm/Group | Fasinumab 1 mg
Number analyzed (Participants) | 586
Milligrams per Liter (mg/L)
  Week 0 | 0.000155 (0.002)
  Week 4: number analyzed (Participants) | 570
  Week 4 | 0.0469 (0.0179)
  Week 8: number analyzed (Participants) | 543
  Week 8 | 0.0644 (0.0275)
  Week 16: number analyzed (Participants) | 502
  Week 16 | 0.0738 (0.0380)
  Week 24: number analyzed (Participants) | 465
  Week 24 | 0.0713 (0.0379)
  Week 44: number analyzed (Participants) | 186
  Week 44 | 0.000349 (0.00476)

18. Secondary Outcome: Number of Participants With At-least One Positive Anti-Drug Antibody (ADA) Development
Description: Immunogenicity was characterized by ADA responses & titers. Responses categories: Pre-existing immunoreactivity - ADA positive response at baseline with all post first dose negative results or positive response at baseline with all post first dose ADA responses < 9-fold over baseline titer levels; Treatment-boosted response - positive response in the assay post first dose, >= 9-fold over baseline titer levels, when baseline results are positive; Treatment-emergent response - ADA positive response post first dose when baseline results = negative or missing.
Time Frame: Baseline up to Week 44
Population: This outcome measure examined only placebo, NSAIDs vs. fasinumab 1mg arms. The ADA analysis set included all participants who received any study drug and had at least 1 non-missing ADA result following the first dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NSAIDs | Fasinumab 1 mg
Number analyzed (Participants) | 291 | 568 | 569
Participants
  Pre-Existing Immunoreactivity | 10 | 9 | 15
  Treated-Boosted Response | 0 | 0 | 0
  Treatment-Emergent Response | 3 | 1 | 4

ADVERSE EVENTS:
Time Frame: First dose to week 44
Groups:
- Fasinumab 1mg Q4W: Participants received SC injection of Fasinumab at a dose of 1 mg Q4W up to 24 weeks and NSAID-matching placebo oral, BID
- Fasinumab 3mg Q4W: Participants received SC injection of Fasinumab at a dose of 3 mg Q4W up to 24 weeks and NSAID-matching placebo oral, BID
- Fasinumab 6mg Q8W: Participants received SC injection of Fasinumab at a dose of 6 mg Q8W up to 24 weeks, alternating with Q8W placebo injections. Participants received placebo injections at the Q4W study visits where study drug was not administered and NSAID-matching placebo oral, BID
Arm/Group | Placebo | NSAIDs | Fasinumab 1mg Q4W | Fasinumab 3mg Q4W | Fasinumab 6mg Q8W
All-Cause Mortality (participants affected / at risk) | 1/309 | 3/609 | 1/609 | 0/58 | 0/59
Serious Adverse Events (participants affected / at risk) | 20/309 | 45/609 | 35/609 | 5/58 | 2/59
Other Adverse Events (participants affected / at risk) | 121/309 | 263/609 | 261/609 | 17/58 | 15/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=309) | NSAIDs (N=609) | Fasinumab 1mg Q4W (N=609) | Fasinumab 3mg Q4W (N=58) | Fasinumab 6mg Q8W (N=59)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6) | 1 (1) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 8 (9) | 2 (2) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device loosening (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 4 (4) | 2 (3) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subchondral insufficiency fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudostroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=309) | NSAIDs (N=609) | Fasinumab 1mg Q4W (N=609) | Fasinumab 3mg Q4W (N=58) | Fasinumab 6mg Q8W (N=59)
Headache (Nervous system disorders) | 48 (113) | 107 (210) | 95 (224) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 25 (29) | 35 (39) | 50 (57) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 22 (26) | 38 (44) | 29 (35) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 (53) | 78 (102) | 82 (109) | 4 (7) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (17) | 44 (60) | 46 (51) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 15 (18) | 30 (31) | 30 (33) | 3 (3) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 5 (5) | 5 (5) | 3 (3) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 5 (5) | 0 (0) | 3 (3)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 6 (7) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT03304379/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT03304379/SAP_001.pdf